CLINICAL TRIAL: NCT06047353
Title: Community Health Advocates for Motivating PAP Use in Our Neighborhoods.
Acronym: Champion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Naresh Punjabi, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20211138; P50MD017347 (NIH)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Motivational Enhancement Therapy (MET) (Experimental): Participants in this group will receive intervention with MET along with PAP therapy. Participants will be in this group for approximately 3 months.
  Interventions: Behavioral: Motivational Enhancement Therapy; Device: Positive Airway Pressure (PAP) therapy
- PAP therapy (Active Comparator): Participants in this group will receive PAP therapy which is the standard of care. Participants will be in this group for approximately 3 months.
  Interventions: Device: Positive Airway Pressure (PAP) therapy

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — Motivational Enhancement Therapy (MET) is based on the principles of motivational interviewing and is designed to promote self-efficacy and maximize behavioral change. MET will be given via phone and/or in person (approximately 30 minutes) at baseline, week 1, week 2, week 4, and week 8.
  Arms: Motivational Enhancement Therapy (MET)
Device: Positive Airway Pressure (PAP) therapy — Positive Airway Pressure (PAP) therapy will be administered as per standard of care.

SUMMARY:
The purpose of this research is to compare the impact of motivational enhancement therapy (MET), delivered by culturally congruent community health care workers (CHWs) versus usual care patients with previously untreated moderate-to-severe obstructive sleep apnea (OSA) on adherence to positive airway pressure (PAP) therapy.

ELIGIBILITY:
Inclusion Criteria

* ≥ 18 years of age
* Moderate-to-severe OSA
* Available to attend study visits and sessions
* Reliable access to a phone

Exclusion Criteria

* Prior or current use of PAP therapy or other treatment (e.g., oral appliance) for OSA
* History of upper airway surgery for OSA
* Moderate to severe insomnia
* Commercial drivers
* Use of non-standard PAP including adaptive servo-ventilation or bi-level positive airway pressure
* Report of motor vehicle accident or near-miss due to sleepiness within the 2 previous years
* Unstable medical conditions that may preclude enrollment in the protocol such as: uncontrolled angina and/or congestive heart failure, uncontrolled blood pressure or resistant hypertension, severe chronic obstructive pulmonary disease, cancer, and active psychiatric disease (e.g., major depression)
* Other sleep disorders (e.g., circadian rhythm disorder)
* Use of supplemental oxygen during wakefulness or sleep
* Central sleep apnea, obesity hypoventilation syndrome or Cheyne-Stokes respiration based on the home sleep apnea test
* Resting awake oxygen saturation (SpO2) < 90%
* Participation in another clinical trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of hours patient adhered to PAP therapy | 3 months
  Measured in the number of hours of use of PAP therapy

SECONDARY OUTCOMES:
Blood pressure | 3 months
  Clinic blood pressure measured in mmHg
Mean Glucose Level | 3 months
  Mean glucose from continuous glucose monitoring measured in mg/dl
Epworth Sleepiness Scale Score | 3 months
  Mean Epworth Sleepiness Score (minimum 1; maximum 24) with higher scores indicating increased sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Punjabi, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No